CLINICAL TRIAL: NCT04760535
Title: Effectiveness of Aligners Versus Rapid Maxillary Expansion on 3D Palatal Volume in Mixed Dentition Patients: a Randomized Controlled Trial
Brief Title: Effectiveness of Aligners Versus Rapid Maxillary Expansion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Turin, Italy (Other)
Responsible Party: Principal Investigator, Tommaso Castroflorio, Aggregate Professor of Orthodontics, University of Turin, Italy
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Maxillary Expansion
Record Dates: First submitted 2021-02-14; First posted 2021-02-18 (Actual); Last update posted 2022-05-25 (Actual); Status verified 2022-05

CONDITIONS: Maxillary Transverse Deficiency (MTD)

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A: Invisalign® First clear aligners (Experimental): The Invisalign® First aligners are fabricated in a multilayer aromatic thermoplastic polyurethane/co-polyester 0.75mm (.030")-thick with a fine 3D manufacturing process.
  Interventions: Device: Invisalign® First Phase I treatment (Align Technology, Inc., Santa Clara, CA, USA)
- Arm B: tooth-borne Hyrax-type maxillary expander (Active Comparator): The Hyrax-type maxillary expander is a tooth-borne expansion appliance that is fixed to the upper second deciduous molars (or to the first permanent molars) using bands and includes a midline 12-mm self-locking screw (Forestadent, Pforzheim, Germany; 0.9 mm, complete turn). The expansion screw is connected to the conventional molar bands or printed clasps, modeled surrounding the molars, via a framework of 0.9mm stainless-steel wire. The framework is soldered to the bands and extending on the palatal side to the deciduous canines. The expander will be fabricated by qualified laboratory technician.
  Interventions: Device: Tooth-borne Hyrax-type maxillary expander

INTERVENTIONS:
Device: Invisalign® First Phase I treatment (Align Technology, Inc., Santa Clara, CA, USA) — Subjects in this arm will be instructed to wear aligners 24h/day for entire duration of the therapy. They will be asked to remove their retainers only while eating, drinking (except water), or cleaning. At the time of appliance delivery, both written and verbal oral hygiene instructions were given, including methods for cleaning appliances themselves. Also, written informed consent were obtained for each patient or the parents.
  Arms: Arm A: Invisalign® First clear aligners
Device: Tooth-borne Hyrax-type maxillary expander — The expansion protocol was one quarter-turn twice a day (0.45 mm activation per day) until overcorrection with the maxillary lingual cusps contacting the mandibular buccal cusps. The expander was left passively for retention for a minimum of 6 months. At the time of appliance delivery, both written and verbal oral hygiene instructions were given, including methods for cleaning appliances themselves. Also, written informed consent were obtained for each patient or the parents.
  Arms: Arm B: tooth-borne Hyrax-type maxillary expander

SUMMARY:
Aim of the study is to assess the effectiveness of Invisalign® First clear aligners compared to tooth-borne Hyrax-type maxillary expander on palatal morphology in growing subjects using 3D technology.

DETAILED DESCRIPTION:
Aim of the study is to assess the effectiveness of Invisalign® First clear aligners compared to tooth-borne Hyrax-type maxillary expander on palatal morphology in growing subjects using 3D technology. This two-arm parallel-group randomized prospective clinical trial will include patients with: indications for maxillary expansion treatment, age between 6 and 10 years old, mixed dentition, good standard of oral hygiene, good compliance during treatment as assessed by the practitioner. Patients will be assigned to one of two expansion methods (arm A: Invisalign® First clear aligners, arm B: tooth-borne Hyrax-type maxillary expander) according to a computer-generated randomization list shortly before the start of expansion Primary outcome measure will be the change in palatal morphology (palatal volume and surface area variations). Secondary outcomes will be: arch dimensions (upper inter-canine width, upper inter-molar width, anterior segment length, posterior segment length), complications, patients' satisfaction and periodontal health. Due to the nature of the intervention blinding will not be possible. Potential statistical differences between the two intervention groups will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* patients who have been diagnosed with transverse maxillary deficiency;
* mixed dentition phase with cervical vertebral maturation stage (CVMS) less than 4;
* fully erupted upper and lower first molars;
* transversal discrepancy ≤5mm
* demonstration of a good standard of oral hygiene (determined through questioning and clinical examination);
* subjects willing to consent to the trial and comply with the trial regime.

Exclusion Criteria:

* any general medical health problems which may influence gingival health, such as those necessitating antibiotic cover as bacteremia prophylaxis, diabetes mellitus, epilepsy, or physical or mental disability;
* permanent teeth extraction-based treatment (third molars excluded);
* morphologic crown anomalies;
* auxiliary treatment during arch expansion stage (such as crossbite elastics);
* posterior interproximal reduction;
* orthognathic surgery treatment planned;
* cleft palate or severe facial deformities.

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2019-01-15 (Actual); Primary Completion 2020-10-15 (Actual); Study Completion 2021-05-03 (Actual)

PRIMARY OUTCOMES:
Palate morphology | 12 months
  The primary outcome will be to evaluate the changes in palatal morphology after the treatment of maxillary deficiencies using two different therapies and to re-evaluate changes over the initial 12-months after the end of the treatment. The changes in palatal morphology are defined as the variation in palatal volume and surface. These will be measured from digitized study models within the boundaries of the palate, the gingival and distal planes, defined as follow. The gingival plane will be created by connecting the midpoints of the dentogingival junction of all upper erupted deciduous and permanent teeth. The distal plane will be created through two points at the distal of the first upper permanent molars perpendicular to the gingival plane.

SECONDARY OUTCOMES:
Upper inter-canine width (ICW) | 12 months
  Upper inter-canine width (ICW) (secondary outcome measure) is the transverse distance between upper canines in millimeters.
Upper inter-molar width (IMW) | 12 months
  Upper inter-molar width (IMW) (secondary outcome measure) is the transverse distance between upper first molars in millimeters.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Turin, Turin, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bruni A, Ferrillo M, Gallo V, Parrini S, Garino F, Castroflorio T, Deregibus A. Efficacy of clear aligners vs rapid palatal expanders on palatal volume and surface area in mixed dentition patients: A randomized controlled trial. Am J Orthod Dentofacial Orthop. 2024 Sep;166(3):203-214. doi: 10.1016/j.ajodo.2024.04.006. Epub 2024 Jul 26. PMID 39066746